CLINICAL TRIAL: NCT01173861
Title: Effectiveness of a Cancer Center Based Physical Activity Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Kristina Karvinen, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 09-0887
Record Dates: First submitted 2010-05-25; First posted 2010-08-02 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer; Quality of Life; Physical Activity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity counseling (Experimental): Group receives face-to-face physical activity counseling.
  Interventions: Behavioral: Physical activity counseling
- Manual (Active Comparator): Group receives physical activity manual.
  Interventions: Behavioral: Physical activity counseling

INTERVENTIONS:
Behavioral: Physical activity counseling — 20-30 minutes of face-to-face physical activity counseling using motivational interviewing followed by 3 20 minute telephone counseling sessions.

SUMMARY:
Purpose: Examine the effectiveness of cancer center-based physical activity counseling on physical activity rates and quality of life in breast cancer survivors.

Hypothesis: Participants in the intervention group will indicate greater step counts and quality of life at the end of the intervention compared to the control group

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer within the last 5 years
* Over the age of 18 years
* female

Exclusion Criteria:

* Non-ambulatory
* Poor cognitive function
* Contraindications for exercise as determined by the PAR-Q

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Effectiveness of a cancer center based physical activity intervention for increasing physical activity in breast cancer survivors. | 8 weeks
  The primary outcome is to examine the effectiveness of a cancer center based physical activity intervention on increasing physical activity as measured by step counts on a pedometer.

SECONDARY OUTCOMES:
Effectiveness of a cancer center based physical activity counseling intervention on increasing quality of life in breast cancer survivors. | 8 weeks
  The secondary outcome is to examine the effectiveness of a cancer center based physical activity counseling intervention on improving quality of life in breast cancer survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina H Karvinen, PhD, Principal Investigator — East Carolina University
Locations (1):
- Leo Jenkins Cancer Center, Greenville, North Carolina, United States